CLINICAL TRIAL: NCT06031090
Title: Intravenous Clonidine Versus Granisetron for Prevention of Post Spinal Anesthesia Shivering in Cesarean Section
Brief Title: Clonidine Versus Granisetron for Shivering Prevension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba M Fathi, Ass. Professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: zu-IRB#10415/26-2-2023
Record Dates: First submitted 2023-08-27; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Post Spinal Anesthesia Shivering
MeSH Terms: interventions — Clonidine; Granisetron; Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: triple blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Cl (clonidine group) (Active Comparator): will be given intravenous Clonidine 0.5 µg/kg diluted in 10ml normal saline 20 minutes before spinal anesthesia
  Interventions: Drug: Clonidine Injection
- Group G (granisetron group) (Active Comparator): will be given intravenous 1mg of granisetron 20 minutes before spinal anesthesia.
  Interventions: Drug: Granisetron Injection
- Group C (control group) (Placebo Comparator): will be given intravenous10ml normal saline 20 minutes before spinal anesthesia
  Interventions: Drug: Normal Saline 10 mL Injection

INTERVENTIONS:
Drug: Clonidine Injection — intravenous Clonidine 0.5 µg/kg diluted in 10ml normal saline 20 minutes before spinal anesthesia
  Arms: Group Cl (clonidine group)
Drug: Granisetron Injection — intravenous 1mg of granisetron diluted in 10ml normal saline 20 minutes before spinal anesthesia.
  Arms: Group G (granisetron group)
Drug: Normal Saline 10 mL Injection — intravenous 10 ml normal saline 20 minutes before spinal anesthesia
  Arms: Group C (control group)

SUMMARY:
Prevention of post spinal anesthesia shivering during cesarean section with its associated discomfort, distress, aggravation of pain, increased metabolic demands, and increased oxygen consumption

DETAILED DESCRIPTION:
Shivering is one of the most important periperative complications seen in clinical practice. Several mechanisms have been postulated for its pathogenesis. Anesthetic-induced inhibition of thermoregulation resulting in hypothermia is an important cause of post anesthesia shivering, uncontrolled spinal reflexes, and cutaneous vasodilation are the other suggested mechanisms involved in the pathogenesis of shivering. Opioid receptors, α2 receptors, and serotonergic receptors also are involved of shivering.

Various drugs were studied for their potential role in prevention of peri-operative shivering such as tramadol, dexmedetomidine, ondansetron, ketamine, and pethidine.

We decided to perform a well-designed study to compare clonidine and granisetron which has been recently introduced as drugs for prevention and control of shivering after spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria: Patient acceptance.,Aged between 21-40 years old, BMI: 18- 30 kg/m2, ASA: I and II., Scheduled for elective cesarean section under spinal anesthesia.

-

Exclusion Criteria:

History of hypersensitivity to drugs used in this study,Patients with history of chronic pain and taking analgesics, Patients with sepsis and Significant cardiac, liver or renal diseases, Uncooperative patients or with psychiatric disorders that prevent surgery under spinal anesthesia, Atrio-ventricular block in any degree, cardiac arrhythmias, valvular heart disease, kidney or liver diseases, neuromuscular disorders and diabetes mellitus

-

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — parturients undergoing cesarean section
Enrollment: 186 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-10-05 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Shivering | Procedure (through out the period of spinal anesthesia)
  • Shivering will be graded according to Tsai and Chu scale (10): 0 = no shivering, 1 = piloerection or peripheral vasoconstriction but no visible shivering, 2 = muscular activity in only one muscle group, 3 = muscular activity in more than one muscle group but not generalized shivering, 4 =shivering involving the whole body

SECONDARY OUTCOMES:
core body temperature | Procedure (preoperative as base and through out the period of spinal anesthesia)
  Core body temperature was detected by measuring tympanic membrane temperature using digital infrared ear thermometer (thermoscan KFT-10; Grnzia, genova, Italy).
Maternal Heart rate | Procedure (preoperative as base and through out the period of spinal anesthesia)
  beats/minute
baby APGAR score | 1 minutes and 5 minutes post natal
maternal blood presure | Procedure (preoperative as base and through out the period of spinal anesthesia)
  mmhg

OTHER OUTCOMES:
maternal oxygen saturation | Procedure (preoperative as base and through out the period of spinal anesthesia)

CONTACTS AND LOCATIONS:
Locations (1):
- Heba M Fathi, Zagazig, Egypt